## The Effect of Interpersonal Relationships and Social Rhythm Therapy Individuals With Bipolar Disorder

Research data were coded with SPSS 22. In the analysis part, firstly, post-hoc analysis will be performed to calculate the power of the sample number, and in treat to analysis will be performed for the validity of randomization. For further analysis of the data, help from an expert statistician will be taken.